CLINICAL TRIAL: NCT05645770
Title: Prospective Memory and Cardiac Activity in Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Chung Cheng University (Other)
Responsible Party: Sponsor
Other Study IDs: 202107146RINB
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: CAD, Prospective Memory
MeSH Terms: interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coronary artery disease
  Interventions: Combination Product: ECG, computerized task
- control
  Interventions: Combination Product: ECG, computerized task

INTERVENTIONS:
Combination Product: ECG, computerized task — ECG for cardiac waves computerized task for prospective memory

SUMMARY:
Previous studies demonstrated an association between cognitive deficit and coronary artery disease (CAD; Abete et al., 2014; Deckers et al., 2017) even after controlling for the effects of age and socioeconomic status (Singh-Manoux et al., 2003). A selective, non-amnestic cognitive impairment profile has also been observed in this patient group (Roberts et al., 2010), with executive function as the most vulnerable cognitive domain (Rostamian et al., 2015).

Prospective memory and CAD Prospective memory (PM) is another facet of executive function that concerns the realization of an intended action (Kvavilashvili, 1998). In addition to the support from memory system, PM strongly relies on attentional and executive control (Kliegel et al., 2011). For example, the two-stage cue-focused view of PM retrieval (McDaniel et al., 2004) posited the importance of "noticing" an action cue before the associated memory search can be initiated. PM is a clinically relevant psychological construct as the failure has been related to quality of life (Doyle et al., 2012), activities of daily living (Woods et al., 2008) and medication adherence (Zogg et al., 2012).

However, little is known about PM function in CAD. Only Habota et al. (2015) reported significant PM deficit in a small group of chronic heart failure patients (N = 19) as compared to healthy controls (N = 24). Therefore, the first aim of the present study is to examine PM performance in people with CAD as compared to their healthy controls.

Prospective memory and cardiac function The association between the brain and the heart has long been recognized (Samuels, 2007). However, the mechanism of cognitive impairment in CAD has not been clearly understood. Researchers proposed several contributing pathological routes including increased platelet activity, thrombo-embolic mechanisms or cardiac output reduction (Abete et al., 2014). The neurovisceral integration model (Smith et al., 2017) proposed a hierarchy of vagal control from intra-cardiac and cardiovascular reactions to representation of multimodal prior expectations that involve the cerebral executive control network. Accumulating evidence supported this notion by demonstrating the link between autonomic nervous system (ANS) and behavioral performance, such as the association between heart rate variability (HRV) and cognitive functions (Forte et al., 2019) and its moderating effect of resting pre-ejection time (PEP; Giuliano et al., 2017).

Few studies investigated the relationship between autonomic responses and PM. Kliegel et al. (2007) and Rothen et al. (2014) verified that there was an association between increased skin conductance responses (SCRs) and the noticing of PM cues in young adults. More recently, Umeda et al. (2016) found that PM performance was associated with an increase in heart rate upon target presentation and with better interoceptive accuracy in college students. They hypothesized that PM was regulated by cardiac afferent signals that facilitate saliency detection and intention retrieval, which was also mediated by interoceptive accuracy. These preliminary findings suggest close relationship between PM and autonomic functions and provide another aspect of the evidence on the brain-heart connection.

However, the methodology adopted in these studies suffered from crude, indirect measures of ANS activity. It is also unclear if the autonomic nervous function compromised by CAD (Montano et al., 2009) would play a role in PM deficit. Hence, the second aim of the present study is to investigate the relationship between PM and cardiac function as measured by HF-HRV (the parasympathetic component) and PEP (the sympathetic component).

ELIGIBILITY:
Inclusion Criteria:

* (1) coronary artery disease noted by coronary angiogram or vascular computer tomography; (2) a history of percutaneous coronary intervention or coronary artery bypass surgery; (3) a history of myocardial infarction or unstable angina; (4) positive exercise electrocardiogram for myocardial ischemia; (5) positive stress radionuclide perfusion scan for myocardial ischemia or infarction; or (6) positive stress cardiac echography for myocardial ischemia.

Exclusion Criteria:

* stroke history, diagnosis of major psychiatric or neurological disorders (such as dementia, major depression, and traumatic brain injury), severe hearing or visual impairment, and movement disturbances.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The CAD group will be recruited from National Taiwan University Hospital Yunlin Branch. Written informed consent will be obtained before entering the study.
  Healthy controls will be recruited from neighboring communities, families of the patients or volunteers in the hospital. Matching procedure will consider age, education, and gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-09 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
PM function in CAD and the relationship of PM performance with parasympathetic and sympathetic measures of cardiac function. | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Douliu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided